CLINICAL TRIAL: NCT00699218
Title: A Pilot Study on Repetitive Transcranial Magnetic Stimulation (rTMS) for Treatment of Bipolar Depression
Brief Title: A Pilot Study on Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment of Bipolar Depression
Acronym: TMS-BD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 200715749
Record Dates: First submitted 2008-06-04; First posted 2008-06-17 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2017-10

CONDITIONS: Mood Disorder; Bipolar Disorder; Major Depression; Depression
Keywords: Bipolar; Depression; TMS; repetitive Transcranial Magnetic Stimulation; treatment; Efficacy; Safety
MeSH Terms: conditions — Mood Disorders; Bipolar Disorder; Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rTMS treatment (Experimental): Active rTMS treatment. Transcranial magnetic stimulation using a device called MagStim
  Interventions: Device: Magnetic Stimulator Rapid2 made by Magstim Company Ltd. U.K.

INTERVENTIONS:
Device: Magnetic Stimulator Rapid2 made by Magstim Company Ltd. U.K. — High frequency repetitive TMS given daily on weekdays for 3 weeks
  Other Names: Repetitive Transcranial Magnetic Stimulation (rTMS)

SUMMARY:
This is a pilot project to study if repetitive Transcranial Magnetic Stimulation (rTMS) will benefit patients with bipolar depression safely. Based on published studies, this study hypothesizes that rTMS on the left dorsal prefrontal lobe will improve symptoms in some patients who have failed at least two medications.

DETAILED DESCRIPTION:
Candidate with bipolar depression will be screened after signing informed consent. Those who meet the selection criteria will be treated with daily rTMS for 3 weeks and be followed-up at 2 weeks. Participants will keep their ongoing medication unless a medication significantly increases the possibility of seizure. They must be on the same dose of antidepressant medication for least 4 weeks without improvement of symptoms before being recruited into the study. Mood and other observed mental status will be measured by standard psychological scales.

ELIGIBILITY:
Inclusion Criteria:

* bipolar I or II patients, currently in a depression episode
* Patient must have failed at least 2 medication
* Score of 21-item Hamilton Rating Scale for Depression (HAM-D)

Exclusion Criteria:

* Rapid cycling bipolar or mixed episode of mood disorder by definition of current DSM criteria
* Substantial risk of suicide during the screening period that requires inpatient care
* Presence of psychosis
* Dual diagnosis of other primary, currently clinically significant severe mental disorders
* History of other significant neurological diseases, such as seizure disorder, stroke, brain tumors, abnormalities in the blood vessels in brain, dementia, Parkinson's disease, Huntington's chorea or multiple sclerosis
* History of any medical event that may increase the risk of having seizure, such as head trauma with unconsciousness for more than 5 minutes or a family history of seizure
* Significant medical complications that may deteriorate during the trial or have increased likelihood of danger consequences
* Patients who are pregnant or intend to become pregnant during the study period
* Any metallic prosthesis in head, neck or upper body (including cardiac pace maker) that cannot be safely removed during treatment
* Current Vagus Nerve Stimulation (VNS) treatment or Electroconvulsive Therapy (ECT) treatment, or with history of failed ECT treatment
* Patient's Motor Threshold for TMS cannot be detected
* Significant side effects which are intolerable during the screening or any later stage of the trial
* Started psychotherapy within the previous 8 weeks or foreseeable psychotherapy will be started or changed in 6 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Xia, M.D., Ph.D., Principal Investigator — Department of Psychiatry and Behavioral Sciences, UC Davis
Locations (1):
- Center for Mind and Brain, Davis, California, United States

REFERENCES:
- See also: PI facilitation — http://www.ucdmc.ucdavis.edu/psychiatry/
- See also: Trial Location: Center for Mind and Brain — http://mindbrain.ucdavis.edu/
- See also: Dr. Xia's blog briefly introducing the trial — http://tms-bd.blogspot.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Active rTMS treatment
  Magnetic Stimulator Rapid2 made by Magstim Company Ltd. U.K.: High frequency repetitive TMS given daily on weekdays for 3 weeks
Period: Overall Study
Arm/Group | Experimental
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 12
Age, Continuous [Mean (Full Range); unit: years] | 50 [19 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (HAM-D)
Description: Scored Questionnaire 0-52, A score of 0-7 is considered to be normal. Scores of 20 or higher indicate moderate, severe, or very severe depression. The higher score means more severe depression.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 15
units on a scale
  Week 1 | 18.4 (8.7)
  Week 2 | 13.4 (6.8)
  Week 3 | 12.4 (6.8)
  Week 5 | 13.7 (7.4)

2. Secondary Outcome: Inventory of Depressive Symptomatology
Description: Self reported depression scale range 0-84. Questionnaire administered at 1,2, and 3 weeks (end of treatment). We also did a 5 week follow-up. The higher scores indicate greater or more severe depression.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 15
units on a scale
  Week 1 | 41.1 (10.2)
  Week 2 | 34.3 (15.5)
  Week 3 | 30.5 (16.1)
  Week 5 | 31.9 (15.2)

ADVERSE EVENTS:
Groups:
- rTMS Treatment: Active rTMS treatment
  Magnetic Stimulator Rapid2 made by Magstim Company Ltd. U.K.: High frequency repetitive TMS given daily on weekdays for 3 weeks
Arm/Group | rTMS Treatment
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 3/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rTMS Treatment (N=15)
Mild Focal Pain (Skin and subcutaneous tissue disorders) | 3 — Discomfort to mild pain in skin area where simulation was applied

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes